CLINICAL TRIAL: NCT00927290
Title: ANRS HC 22, PEGLIST-C, Multicenter, Randomized Controlled Trial of Pioglitazone vs. Placebo in Association With Pegylated Interferon and Ribavirin in Patients With Chronic Hepatitis C, Non 2 or 3 Genotypes and Insulin Resistance
Brief Title: Pioglitazone vs. Placebo in Association With Pegylated Interferon and Ribavirin in HCV Patients With Insulin Resistance
Acronym: PEGLIST C
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Suspension of use of medicine containing Pioglitazone by French regulatory agency
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-006225-14
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Hepatitis C; Insulin Resistance
Keywords: hepatitis C; insulin resistance; glitazones; pioglitazone; steatosis; viral kinetics; antiviral response
MeSH Terms: conditions — Hepatitis C, Chronic; Insulin Resistance; Hepatitis C; Fatty Liver | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Pioglitazone, 16 weeks before and during antiviral combination therapy
  Interventions: Drug: Pioglitazone
- 2 (Placebo Comparator): Pioglitazone placebo, 16 weeks before and during antiviral combination therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone, 45 mg QD (30 mg QD the first month)
  Arms: 1
Drug: Placebo — Placebo 45 mg QD (30 mg QD the first month)
  Arms: 2

SUMMARY:
The purpose of this study is to test whether the correction of insulin resistance with pioglitazone, will improve the response to antiviral treatment.

DETAILED DESCRIPTION:
In patients infected with genotypes 1, 4, 5 and 6, the response rate to antiviral therapy remains suboptimal (less than one in two patients have a sustained virological response), which justifies the search for strategies optimizing the results of antiviral therapy. Some factors associated with non response have been identified. Among the modifiable factors, numerous series have shown that insulin resistance adversely impacts the rate of sustained virological response. The aim of this study is to determine whether the pharmacological correction of insulin resistance through therapy with glitazones restores higher rates of viral eradication and to determine the impact on the kinetics of viral response. Patients will be randomized to receive pioglitazone or placebo starting 4 months before initiating pegylated interferon and ribavirin and continued throughout the whole antiviral treatment period.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Chronic HCV infection documented by PCR with genotype HCV-1, 4, 5 or 6
* Naive Patient(never treated with antivirals for HCV)
* HOMA score higher than 2.5
* Patient for which the investigator decided to start antiviral treatment for chronic hepatitis C

Exclusion Criteria:

* Cardiovascular disease: heart failure stage NYHA II, III or IV, unstable angina, myocardial infarction in the previous year, cardiac surgery or stroke
* Alcohol consumption exceeding 40 g / day
* Decompensated liver disease: Child-Pugh B 8 or higher, or one of the following : bilirubin over 35 mol / L, TP below 50%, ascites, encephalopathy
* Hepatocellular carcinoma or any other neoplasm (except if in remission for > 5 years)
* Other documented chronic liver disease
* Insulin treated diabetes
* HBV or HIV co-infection infection confirmed
* Thrombocytopenia below 50 000/mm ³; neutropenia below 750/mm ³ or hemoglobin below 11 g / dL
* Drug-induced steatosis(tamoxifen, glucocorticosteroids, amiodarone, tetracyclines).
* Bone marrow or solid organ transplantation
* Pregnancy or breastfeeding, or desire for pregnancy during the study period.
* Patients under legal protection or unable to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-12-03 (Actual); Primary Completion 2012-07-06 (Actual); Study Completion 2012-07-06 (Actual)

PRIMARY OUTCOMES:
Decrease in the HOMA score below 2 after 4 months of treatment with pioglitazone or placebo(at W16). The efficiency is defined as a higher proportion of subjects with HOMA <2 in the pioglitazone group than in the group treated with placebo pioglitazone. | W16

SECONDARY OUTCOMES:
Kinetics of decrease in viral response to pegylated interferon. Early virological response rates. Rates of sustained virological response. Effect on steatosis | EVR at W16 and W28 SVR at W88

CONTACTS AND LOCATIONS:
Overall Officials: Vlad RATZIU, MD, PHD, Principal Investigator — Hôpital Pitié--Salpêtrière, 83 Bd de l'Hôpital 75651 Paris cedex 13, FRANCE
Locations (1):
- Hôpital Pitié Salpêtrière, Service d'hépatogastroentérologie, Paris, France